CLINICAL TRIAL: NCT05595824
Title: Open Multicenter Study for Assessment of Efficacy and Safety of the Drug JCBC00101, Capsules (PROMOMED RUS LLC, Russia) in Relation to COVID-19 in Adult Population
Brief Title: Open Multicenter Study for Assessment of Efficacy and Safety of Molnupiravir in Adult Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Promomed, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOL-112021
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Molnupiravir; Esperavir
MeSH Terms: conditions — COVID-19 | interventions — molnupiravir; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JCBC00101 (Molnupiravir, Esperavir) (Experimental): Group 1 (n=120) received the study drug JCBC00101, capsules 800 mg, 2 times a day with 12 ±2 hours interval for 5 days in the setting of pathogenetic and symptomatic therapy provided by Interim Guidelines for the prevention, diagnosis and treatment of COVID-19 approved by the Russian Ministry of Health (version 14, December 27, 2021) or valid as of the time of the study
  Interventions: Drug: Molnupiravir (Esperavir)
- Standard of care (Active Comparator): Group 2 (n=120) patients receive standard therapy prescribed in accordance with the recommended treatment regimens included in the Interim Guidelines for the prevention, diagnosis and treatment of COVID-19 approved by the Russian Ministry of Health (version 14, December 27, 2021) or valid as of the time of the study by decision of the investigator and taking into accountthe availability of drugs at the study site (Favipiravir, Umifenovir, IFN α, used incombination with each other).
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Molnupiravir (Esperavir) — Capsules 800 mg, 2 times a day with 12 ±2 hours interval for 5 days
  Other Names: JCBC00101
  Arms: JCBC00101 (Molnupiravir, Esperavir)
Drug: Standard of care — The administration of 'Standard of care' drugs was done according to the regimen recommended in the 'COVID-19 TreatmentGuidelines'(Version 14 of 27.12.2021), or inforce at the time of the study
  Arms: Standard of care

SUMMARY:
This is open-labe randomized multicenter comparative Phase III study conducted in 12 medical facilities. The objective of the study is to evaluate efficacy and safety of the drug JCBC00101, capsules in the setting of pathogenetic and symptomatic therapy as compared to standard therapy in outpatients with COVID-19.

DETAILED DESCRIPTION:
Upon signing the informed consent form and screening, 240 eligible outpatients with mild or moderate COVID-19 were randomized at a 1:1 ratio to receive either molnupiravir capsules, 800 mg, 2 times a day with 12 ±2 hours interval for 5 days, or SOC

ELIGIBILITY:
Inclusion Criteria:

1. Availability of PIS Informed Consent Form signed and dated by a patient.
2. Male and female subjects aged 18 to 80 inclusive as of the time of signing the PIS Informed Consent Form.
3. Confirmed COVID-19 at screening stage: positive for SARS-CoV-2 RNA laboratory test with nucleic acid amplification techniques (NAAT) or SARS-CoV-2 antigen with immunochromatographic assay.

   SARS-CoV-2 test results obtained up to 5 days prior to randomization may be taken into account upon availability of supporting documentation.
4. Mild or moderate SARS-CoV-2 induced infection.
5. At least one of the following COVID-19 symptoms as of the time of screening and randomization: nasal congestion or rhinitis; sore throat; dyspnoea or respiratory distress on exertion; cough; tiredness; pain in muscles or throughout the body; headache; chills; fever (body temperature >38 ⁰С); nausea; vomiting; diarrhea; anosmia; ageusia.
6. Disease onset (first symptom) within not more than 5 days prior to randomization .
7. The patient agrees and is able to take oral drug products.
8. Patient's consent to use reliable contraception methods during the entire study and for 3 weeks after the end of the study. Reliable contraception methods are: sexual abstinence, the use of a condom combined with a spermicidal agent.

Female subjects incapable of bearing children (history: hysterectomy, tubal ligation, infertility, menopause for more than 2 years), as well as male subjects with infertility or a history of vasectomy may participate in the study.

Exclusion Criteria:

1. Hypersensitivity to the study drug components.
2. Favipiravir intake within 7 days prior to screening.
3. Necessity to use drugs included the prohibited therapy list.
4. Hospitalization necessity or expected hospitalization due to COVID-19 within 48 hrs after randomization.
5. Severe and extremely severe disease signs as of the time of screening.
6. Vaccination within less than 4 weeks prior to screening.
7. Possible or confirmed moderate COVID-19 within 6 months prior to screening.
8. Possible or confirmed history of severe or very severe COVID-19.
9. Patients with chronic kidney disease on dialysis or with GFR < 30 mL/min as of the time of screening.
10. History of HIV, syphilis, HBV and/or HCV.
11. Blood components transfusion within 7 days prior to screening.
12. Alcohol, pharmacological and/or drug dependence (history and/or at the time of screening).
13. Schizophrenia, schizoaffective disorder, bipolar disorder, or other psychiatric disorder (history or suspected) at the time of screening.
14. Any history data that may complicate, in the opinion of the investigator, interpretation of the study results or create additional risk for the patient due to his/her participation in the study.
15. Unwillingness or inability of a patient to comply with the Protocol procedures (in the opinion of the investigator).
16. Pregnant or lactating women, or women planning a pregnancy.
17. Participation in another clinical study within 3 months prior to enrollment in the present study.
18. Other conditions investigator considers as preventing the patient from inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of patients with COVID-19 severity increase as compared from baseline to Visit 4. | From baseline to Visit 4 (days 14-15)
  Patient severity score at screening and during treatment was determined as per Current clinical Guidelines, version 14 (December 27,2021).

SECONDARY OUTCOMES:
Clinical status changes as per the categorical ordinal clinical improvement WHO scale | From baseline to Visit 2 (days 6-7), 3 (days 11-12), 4 (days 14-15), 5 (days 21±1), 6 (study completion, day 28±1)
  The score as per the categorical ordinal clinical improvement WHO scale
Clinical status deterioration incidence as per the categorical ordinal clinical improvement WHO scale by ≥ 1 category | From baseline to Visit 2 (days 6-7), 3 (days 11-12), 4 (days 14-15)
  The proportion of patients with clinical status deterioration as per the categorical ordinal clinical improvement scale of ≥ 1 category
Prevalence of patients with category 0 as per categorical ordinal clinical improvement WHO scale | From baseline to Visit 2 (days 6-7), 3 (days 11-12), 4 (days 14-15)
  The proportion of patients with category 0 as per the categorical ordinal clinical improvement scale
Prevalence of patients with category 1 and less according to clinical improvement WHO scale | From baseline to Visit 2 (days 6-7), 3 (days 11-12), 4 (days 14-15)
  The proportion of patients with category 1 and less as per the categorical ordinal clinical improvement scale
Prevalence of patients with negative SARS-CoV-2 RNA test | From baseline to Visit 2 (days 6-7), 3 (days 11-12), 4 (days 14-15)
  The proportion of patients with negative SARS-CoV-2 RNA test
Symptoms intensity score as per COVID-19 Major Symptom Rating Scale. | From baseline to Visit 2 (days 6-7), 3 (days 11-12), 4 (days 14-15), 5 (days 21±1), 6 (study completion, day 28±1)
  The proportion of patients with Symptoms intensity score as per COVID-19 Major Symptom Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy Pushkar, Academician, Principal Investigator — Moscow State Clinical Hospital №50
Locations (12):
- Russia (12):
  - Regional Budget Healthcare Institution "Ivanovo clinical hospital", Ivanovo
  - Kirov State Medical University of Ministry of Health of the Russian Federation, Kirov
  - State Budgetary Healthcare Institution City Clinical Hospital named after S. I. Spasokukotskiy of Moscow Healthcare Department, Moscow
  - Professorskaya klinika, LLC, Perm
  - Ryazan State Medical University named after academician I.P. Pavlov of Ministry of Health of the Russian Federation, Ryazan
  - Avrora MedFort, LLC, Saint Petersburg
  - OrCli Hospital, LLC, Saint Petersburg
  - Ogarev Mordova State University of Ministry of Health of the Russian Federation, Saransk
  - Regional State Budget Healthcare Institution "Clinical hospital No. 1", Smolensk
  - Smolensk State Medical University of Ministry of Health of the Russian Federation, Smolensk
  - Uromed, LLC, Smolensk
  - State Budgetary Healthcare Institution of Yaroslavl Region "Clinical hospital No. 3", Yaroslavl

IPD SHARING:
Plan to Share IPD: No